CLINICAL TRIAL: NCT04663958
Title: Predictive Value of Ariscat Risk Index In The Development of Postoperative Pulmonary Complication After Major Abdominal Cancer Surgery
Brief Title: Predictive Value of Ariscat Index In The Development of Pulmonary Complication After Major Abdominal Cancer Surgery
Status: Completed | Type: Observational
Sponsor: Dr Abdurrahman Yurtaslan Ankara Oncology Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Mustafa Kemal ŞAHİN, Principal Investigator, Dr Abdurrahman Yurtaslan Ankara Oncology Training and Research Hospital
Other Study IDs: 2019-11/459
Record Dates: First submitted 2020-11-24; First posted 2020-12-11 (Actual); Last update posted 2022-11-18 (Actual); Status verified 2022-11

CONDITIONS: Postoperative Complications; Cancer; Pulmonary Complication; Atelectasis; Abdominal Surgery; Pneumonia
MeSH Terms: conditions — Postoperative Complications; Neoplasms; Pulmonary Atelectasis; Pneumonia | interventions — Mass Screening

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Detection / Screening — The patients were followed up in the postoperative care unit. The presence of postoperative pulmonary complications was evaluated, and the time of discharge was recorded. On the 30th day after discharge, patients were called and checked their status in terms of mortality.

SUMMARY:
The term postoperative pulmonary complication is the development of any complications affecting the respiratory system after anesthetic and surgery procedures. The ARISCAT risk assessment score is a seven-variable regression model that divides patients into low, moderate, and high-risk groups. In this study, the investigators aimed to investigate the effectiveness of the ARISCAT risk scoring index in predicting postoperative pulmonary complication development in patients scheduled for major abdominal cancer surgery.

DETAILED DESCRIPTION:
Postoperative pulmonary complications (PPC) are one of the major causes of postoperative morbidity and mortality. Mortality and morbidity are 14-30% in patients with PPC, while it is 0.2-3% in patients without PPC. Its incidence is variable (<1% to 19%) and is more common than cardiac complications. Unfortunately, PPCs prolong the hospital stay significantly (up to 13-17 days), which means postoperative delirium, infection, and cost increase. The causes of PPCs are varied, and their physiopathology is well explained [3]. However, the rate of risk identification and scoring is not known. The synergistic effects of the patient's medical condition, general anesthesia, and surgery type on the respiratory system complicate the problem.The surgical approach, anesthesia method, and preoperative risk factors of the patients play an important role in the development of PPC.

This study was conducted after the approval from Dr. Abdurrahman Yurtaslan Oncology SUAM Ethics Committee in Ankara, Turkey (Between December 2020 - July 2021) (Ethics Committee Decision No: 2019-11 / 459). After informing all the patients included in the study, verbal and written consent were obtained. 410 patients over 18 years of age, who were scheduled for general anesthesia and whose ASA physical score was 1-4, were included in the study.

Demographic data of the patients, preoperative antibiotic prophylaxis, chronic diseases, ASA scores, preoperative hemoglobulin values, functional status, history of pulmonary system disease in the last 30 days, history of smoking and the amount of cigarette consumption, history of steroid use, chemotherapy and radiotherapy history, anesthesia method, surgical incision side (lower-upper abdominal), premedication status, intraoperative ventilation parameters (tidal volume, PEEP, peak pressure, fiO2 ratio), pneumoperitoneum pressure, amount of colloid / crystalloid product used, erythrocyte suspension and amount used, laparoscopic or open surgery, emergency or elective surgery, the duration of operation, and postoperative analgesia method (such as intravenous or epidural patient-controlled analgesia) were recorded. The ARISCAT risk assessment scores of the patients were also evaluated and recorded preoperatively.

The patients were followed up in the postoperative care unit. The presence of postoperative pulmonary complications was evaluated, and the time of discharge was recorded. On the 30th day after discharge, patients were called and checked their status in terms of mortality. Postoperative pulmonary complications were defined by the development of one of the following new findings. The European Perioperative Clinical Outcome Definitions (EPCO) were used for this definition.

These findings; Respiratory Failure, Respiratory infection, Aspiration Pneumonia, Pleural effusion, Pneumothorax, Atelectasis, Bronchoconstriction, Pneumonia, ARDS, Pulmonary Embolism, Pulmonary Edema, Unplanned emergency re-intubation, Leaving as intubated from the operation room.

ELIGIBILITY:
Inclusion Criteria:

1. Over 18 years of age
2. Who were scheduled for general anesthesia
3. Whose ASA physical score was 1-4

Exclusion Criteria:

1. ASA physical status> 4
2. Pregnant women
3. Intubated patients before the operation
4. Patients who had surgery due to a previous surgical complication
5. Severe cardiovascular disease
6. Severe hemodynamic instability

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A total of 420 patients operated in General Surgery, Urology, and Gynecological Oncology departments were included in the study. Seven of these patients were excluded from the study because they did not sign the written consent, and three patients were excluded due to a lack of data.
Sampling Method: Non-Probability Sample
Enrollment: 410 (Actual)
Dates: Start 2020-12-21 (Actual); Primary Completion 2021-06-18 (Actual); Study Completion 2021-08-18 (Actual)

PRIMARY OUTCOMES:
Effectiveness of the ARISCAT risk scoring index | postoperative first 7 days
  to investigate the effectiveness of the ARISCAT risk scoring index in predicting the development of PPC in patients undergoing major abdominal cancer surgery

SECONDARY OUTCOMES:
Correlation between age (years) and PPC | postoperative first 30 days
  Whether there is a correlation between age (years) and PPC
Correlation between gender(male or female) and PPC | postoperative first 30 days
  Whether there is a correlation between gender (male or female) and PPC
Correlation between BMI (kg/m^2) and PPC | postoperative first 30 days
  Whether there is a correlation between BMI (kg/m^2) and PPC
Correlation between history of smoking and the amount of cigarette consumption level (packs/year) and PPC | postoperative first 30 days
  Whether there is a correlation between smoking level (packs/year) and PPC
Correlation between ASA physical score (1-4) and PPC | postoperative first 30 days
  Whether there is a correlation between ASA physical score (1-4) and PPC
Correlation between Preoperative Sp02(>96%, 91%-95%, <90%) and PPC | postoperative first 30 days
  Whether there is a correlation between Preoperative Sp02(>96%, 91%-95%, <90%) and PPC
Correlation between preoperative hemoglobulin values (gram / deciliter) and PPC | postoperative first 30 days
  Whether there is a correlation between preoperative hemoglobulin values (gram / deciliter) and PPC
Correlation between surgical incision side (lower-upper abdominal) and PPC | postoperative first 30 days
  Whether there is a correlation between surgical incision side (lower-upper abdominal) and PPC
Correlation between laparoscopic or open surgery and PPC | postoperative first 30 days
  Whether there is a correlation between laparoscopic or open surgery and PPC
Correlation between , emergency or elective surgery and PPC | postoperative first 30 days
  Whether there is a correlation between , emergency or elective surgery and PPC
Correlation between the duration of operation (<2 hours, 2-3 hours, more than 3 hours) and PPC | postoperative first 30 days
  Whether there is a correlation between the duration of operation (<2 hours, 2-3 hours, more than 3 hours) and PPC
Correlation between postoperative analgesia method (such as intravenous or epidural patient-controlled analgesia) and PPC | postoperative first 30 days
  Whether there is a correlation between postoperative analgesia method (such as intravenous or epidural patient-controlled analgesia) and PPC

CONTACTS AND LOCATIONS:
Overall Officials: MUSTAFA KEMAL SAHIN, Dr, Study Director — Ankara Oncology Education and Research Hospital Clinic of Anesthesiology and Reanimation
Locations (1):
- Dr. Abdurrahman Yurtaslan Ankara Oncology Education and Research Hospital Clinic of Anesthesiology and Reanimation, Ankara, Yenimahalle, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Canet J, Gallart L, Gomar C, Paluzie G, Valles J, Castillo J, Sabate S, Mazo V, Briones Z, Sanchis J; ARISCAT Group. Prediction of postoperative pulmonary complications in a population-based surgical cohort. Anesthesiology. 2010 Dec;113(6):1338-50. doi: 10.1097/ALN.0b013e3181fc6e0a. PMID 21045639
- [Background] Miskovic A, Lumb AB. Postoperative pulmonary complications. Br J Anaesth. 2017 Mar 1;118(3):317-334. doi: 10.1093/bja/aex002. PMID 28186222
- [Background] Arozullah AM, Khuri SF, Henderson WG, Daley J; Participants in the National Veterans Affairs Surgical Quality Improvement Program. Development and validation of a multifactorial risk index for predicting postoperative pneumonia after major noncardiac surgery. Ann Intern Med. 2001 Nov 20;135(10):847-57. doi: 10.7326/0003-4819-135-10-200111200-00005. PMID 11712875
- [Background] Yang CK, Teng A, Lee DY, Rose K. Pulmonary complications after major abdominal surgery: National Surgical Quality Improvement Program analysis. J Surg Res. 2015 Oct;198(2):441-9. doi: 10.1016/j.jss.2015.03.028. Epub 2015 Mar 18. PMID 25930169
- [Background] Gupta H, Ramanan B, Gupta PK, Fang X, Polich A, Modrykamien A, Schuller D, Morrow LE. Impact of COPD on postoperative outcomes: results from a national database. Chest. 2013 Jun;143(6):1599-1606. doi: 10.1378/chest.12-1499. PMID 23287892
- [Background] Jammer I, Wickboldt N, Sander M, Smith A, Schultz MJ, Pelosi P, Leva B, Rhodes A, Hoeft A, Walder B, Chew MS, Pearse RM; European Society of Anaesthesiology (ESA) and the European Society of Intensive Care Medicine (ESICM); European Society of Anaesthesiology; European Society of Intensive Care Medicine. Standards for definitions and use of outcome measures for clinical effectiveness research in perioperative medicine: European Perioperative Clinical Outcome (EPCO) definitions: a statement from the ESA-ESICM joint taskforce on perioperative outcome measures. Eur J Anaesthesiol. 2015 Feb;32(2):88-105. doi: 10.1097/EJA.0000000000000118. PMID 25058504
- [Background] Perilli V, Aceto P, Ancona P, De Cicco R, Papanice D, Magalini S, Pepe G, Cozza V, Gui D, Lai C, Sollazzi L. Role of surgical setting and patients-related factors in predicting the occurrence of postoperative pulmonary complications after abdominal surgery. Eur Rev Med Pharmacol Sci. 2018 Jan;22(2):547-550. doi: 10.26355/eurrev_201801_14208. PMID 29424916